CLINICAL TRIAL: NCT04070950
Title: Longitudinal Study of the Couple Relationship of Women With Pelvic Cancer: Impact on Sexuality
Brief Title: Sexuality of Women With Pelvic Cancer
Acronym: FECAPSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2008/39
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Sexual Behavior; Pelvic Cancer
MeSH Terms: conditions — Sexual Behavior; Pelvic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Single group: Interview of patients with cancer of the cervix or uterine body, or ovary between the time of diagnosis and 3 months after the end of their last cancer treatment (not the object of the study).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Two self-questionnaires

SUMMARY:
This study aims to study in patients with cancer of the cervix or the body of the uterus, or the ovary between the time of diagnosis and 3 months after the end of the last treatment: the evolution of the relationship of couple, and more particularly of communication (verbal and non-verbal) concerning sexuality, before and during cancer.

DETAILED DESCRIPTION:
The representations associated with sexuality and cancer seem antinomic: wellbeing / death, and yet combine in the experience of cancer. The latter has an impact on sexuality in terms of satisfaction or sexual activity and on the relationship in terms of support.

In addition, various studies show the psychological impact of treatments on the couple's relationship or the body image of women with cancer. Their abilities to seduce are affected and explain the decrease of their sexual activity during the treatments: a communication, valuing the femininity, would it then facilitate the relations of couple? There is no work that considers sexuality in a systematic way (sexual act and verbal and non-verbal communication) and apprehends its link with the evolution of the relationship, from the diagnosis of cancer to the end of treatments.

This study aims to study in patients with cancer of the cervix or the body of the uterus, or the ovary between the time of diagnosis and 3 months after the end of the last treatment: the evolution of the relationship of couple, and more particularly of communication (verbal and non-verbal) concerning sexuality, before and during cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Life in a couple or single with a regular partner for at least 3 months
* Cancer of the cervix or uterine body or ovarian cancer, in first diagnosis and treatment
* Whatever the stage of cancer
* Curative treatment
* Support in one of the participating centers
* Possible follow-up of all stages of the research

Exclusion Criteria:

* Presence of metastases
* History of other cancer
* History of severe psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with cancer of the cervix or uterine body, or ovarian
Study Population: Women with cancer of the cervix or uterine body, or ovarian
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2010-05-20 (Actual); Study Completion 2010-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of sexual activity | 3 months after the end of therapeutic treatment (not the object of the study)
  Questionnaire SAQ : Sexual Activity Questionnaire, contains 21 items divided into three parts: the first part allows to know if a woman is sexually active or not, the second part allows to define the reasons for this activity or its absence. The third part of the questionnaire filled out by sexually active women aims to explore the pleasure generated by sex (desire, satisfaction, frequency), discomfort during intercourse, especially due to vaginal dryness and pain as well as the habits of the patient before the illness.

CONTACTS AND LOCATIONS:
Overall Officials: Alain RAVAUD, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No